CLINICAL TRIAL: NCT01456871
Title: Finger Muscle Reaction After Electrical Stimuli to the Human Finger Pulley System; a Pilot Study
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Richard A. Berger, MD, Mayo Clinic
Other Study IDs: 11-004310
Record Dates: First submitted 2011-10-19; First posted 2011-10-21 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
Keywords: Mechanoreceptors; PIP joint; Ligamento-muscular reflexes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy adult females: Females, aged 20 to 30 with no history of upper extremity injury or disorder in the non-dominant arm, no history of neurologic or bleeding disorder, and no evidence of Linburg-Comstock syndrome.
  Interventions: Procedure: Guided insertion of electrodes; Procedure: Electromyographic (EMG) recording

INTERVENTIONS:
Procedure: Guided insertion of electrodes — Fine-wire needle electrodes (30mm x 27gauge needle with a pairs of 0.051mm, insulated, hooked wires, Motion Lab Systems, Baton Rouge, LA) guided by sonographic evaluation of the pulley system using a Philips iU22 Ultrasound Machine (Philips Ultrasound Systems, Bothell, WA), a 17-5 MHz linear array transducer, and standard ultrasound gel.
Procedure: Electromyographic (EMG) recording — EMG signal recording, performed with an MA 300 EMG system (Motion Lab Systems, Baton Rouge, LA).

SUMMARY:
The purpose of the study is to gain a better understanding of mechanoreceptors in the PIP joint ligamento-muscular reflexes and their role is.

DETAILED DESCRIPTION:
Encapsulated nerve endings called mechanoreceptors are end components of afferent nerves and have specialized end organs surrounding the nerve terminal. Those receptors are concentrated in various human periarticular tissues. It is believed that these mechanoreceptors in the periarticular tissues are related to muscle reflexes. However, it is still unknown which type of mechanoreceptors contribute to the muscle reflexes and whether the mechanoreceptors excite and/or inhibit muscle activation. In the investigators previous studies, mechanoreceptors in the human proximal interphalangeal (PIP) joint and surrounding structures have been extensively examined. The investigators have identified that Pacini-like nerve endings in the PIP joint were found in substantial numbers in the junction of the C1 pulley and accessory collateral ligaments. The investigators hypothesize that the Pacini-like nerve endings in the junction of the C1 pulley generate activity in the associated flexor muscle/tendon in the finger.

ELIGIBILITY:
Inclusion criteria:

- Females aged 20-30

Exclusion criteria:

* A history of any upper extremity injury or disorder in the non-dominant arm
* A history of any neurologic or bleeding disorder, or taking blood-thinning medication.
* Presence of Linbug-Comstock syndrome

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Berger, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States